CLINICAL TRIAL: NCT00412074
Title: Establishing the Vitamin D Requirements During Lactation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Carol Wagner, Professor of Pediatrics, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HD047511; R01HD047511 (NIH)
Record Dates: First submitted 2006-12-13; First posted 2006-12-15 (Estimated); Results first posted 2016-06-03 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Vitamin D Deficiency
Keywords: Breastfeeding; Vitamin D; Vitamin D deficiency
MeSH Terms: conditions — Vitamin D Deficiency; Breast Feeding | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control 400 IU vitamin D3 (Active Comparator): 400 IU vitamin D3/day given to lactating women and 400 IU vitamin D3/day given as oral supplement to infant in dyad
  Interventions: Drug: 400 IU Vitamin D3 (cholecalciferol)
- 2400 IU vitamin D3 (cholecalciferol) (Experimental): 2400 IU vitamin D3 given to lactating mother: 400 IU vitamin D3 from a prenatal vitamin and 2000 IU vitamin D3 and 0 IU vitamin D3 (placebo) given to her breastfeeding infant
  Interventions: Drug: 2400 IU Vitamin D3 (cholecalciferol)
- 6400 IU vitamin D3 (cholecalciferol) (Experimental): 6400 IU vitamin D3 given to lactating mother: 400 IU vitamin D3 from a prenatal vitamin and 6000 IU vitamin D3 and 0 IU vitamin D3 (placebo) given to her breastfeeding infant
  Interventions: Drug: 6400 IU Vitamin D3 (cholecalciferol)

INTERVENTIONS:
Drug: 400 IU Vitamin D3 (cholecalciferol) — 400 IU vitamin D3/day given to lactating mother and 400 IU vitamin D3/day given as oral supplement to her infant
  Arms: Control 400 IU vitamin D3
Drug: 2400 IU Vitamin D3 (cholecalciferol) — 2400 IU vitamin D3/day given to lactating mother and 0 IU vitamin D3/day (placebo) given as oral supplement to her infant
  Arms: 2400 IU vitamin D3 (cholecalciferol)
Drug: 6400 IU Vitamin D3 (cholecalciferol) — 6400 IU vitamin D3/day given to lactating mother and 0 IU vitamin D3/day (placebo) given as oral supplement to her infant
  Arms: 6400 IU vitamin D3 (cholecalciferol)

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of maternal and infant vitamin D supplementation as a function of ethnicity and latitude in the prevention of vitamin D deficiency in the breastfeeding mother-infant pair. The findings of this study will generate important new information for health care professionals and policy makers with regard to vitamin D requirements and the potential benefit to both mother and infant

DETAILED DESCRIPTION:
Mothers from two study sites at different latitudes will be randomized to receive 1 of 3 treatment regimes of vitD3. Mothers, lactating or nonlactating controls will be randomized to either Group A: standard treatment(400 IU D3/d), Group B: (2,400 IU D3/d), or Group C: (6,400 IU D3/d. Infants of mothers randomized to Group A will receive 400 IU D3/d (recommended practice) and infants of mothers assigned to Groups B or C will receive placebo. On 2/5/2009, the protocol was amended and the Group B arm was dropped; infants of active subjects randomized to Group B as of 2/5/2009 were put on open label treatment (400 IU D3/d) through study completion. Newly enrolled subjects after this date were randomized to Group A or Group C only.

By measuring an array of indicators,calcium homeostasis and skeletal remodeling in the postpartum mother and the breastfeeding infant will be monitored. Through this study, the prevalence of vitD deficiency in the breastfeeding dyad and the utility of maternal therapeutic intervention with VitD3 will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Mother plans to breastfeed exclusively for at least six months
* Mother is in good health
* Infant is 35 weeks' gestation or greater
* Breastfeeding infant is in good health ( Level I nursery; or Level II nursery but not requiring oxygen therapy or parenteral nutrition beyond first 72 hours).

Exclusion Criteria:

* Mother does not plan to breastfeed exclusively for the first six months (plans to use formula for infant's feedings during the first six months
* Infant has been admitted to Neonatal Intensive Care unit requiring oxygen therapy or parental nutrition beyond the first 72 hours
* Infant is less than 35 weeks' gestation
* Infant has been diagnosed with a congenital anomaly or abnormal chromosomal pattern
* Mother has a history of endocrine dysfunction involving parathyroid gland, diabetes, or calcium abnormalities related to renal disease such that calcium parameters are abnormal
* Mother has history of hypercalciuria

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 460 (Actual)
Dates: Start 2006-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce W. Hollis, Ph.D, Principal Investigator — Medical University of South Carolina; Carol L. Wagner, MD, Principal Investigator — Medical University of South Carolina; Thomas C. Hulsey, Ph.D, Study Chair — Medical University of South Carolina
Locations (2):
- United States (2):
  - University of Rochester Medical Center, Rochester, New York
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Derived] Ramadurai S, Andrews C, Cheema S, Thomas R, Wagner CL, Sen S. Maternal Predictors of Breast Milk Plasmalogens and Associations with Infant Body Composition and Neurodevelopment. Clin Ther. 2022 Jul;44(7):998-1009. doi: 10.1016/j.clinthera.2022.06.003. Epub 2022 Jul 29. PMID 35909001
- [Derived] Andrews L, Phlegar K, Baatz JE, Ebeling MD, Shary JR, Gregoski MJ, Howard CR, Hollis BW, Wagner CL. Comparison of Infant Bone Mineral Content and Density After Infant Daily Oral Vit D 400 IU Supplementation Versus Nursing Mother Oral 6,400 IU Supplementation: A Randomized Controlled Lactation Study. Breastfeed Med. 2022 Jun;17(6):493-500. doi: 10.1089/bfm.2021.0281. Epub 2022 Mar 10. PMID 35271380
- [Derived] Pouch GG, Ebeling M, Shary JR, Hollis BW, Howard CR, Wagner CL. Evaluating Vitamin D Status in Infants Less than Seven Months; What Are the Preferred Biochemical Measurements? Breastfeed Med. 2022 May;17(5):422-428. doi: 10.1089/bfm.2021.0237. Epub 2022 Feb 23. PMID 35196139
- [Derived] Wagner CL, Hulsey TC, Ebeling M, Shary JR, Asghari G, Howard CR, Baatz JE, Newton DA, Wahlquist AE, Reed SG, Taylor SN, Lawrence RA, Hollis BW. Safety Aspects of a Randomized Clinical Trial of Maternal and Infant Vitamin D Supplementation by Feeding Type Through 7 Months Postpartum. Breastfeed Med. 2020 Dec;15(12):765-775. doi: 10.1089/bfm.2020.0056. Epub 2020 Sep 11. PMID 32915638
- [Derived] Bell KA, Wagner CL, Perng W, Feldman HA, Shypailo RJ, Belfort MB. Validity of Body Mass Index as a Measure of Adiposity in Infancy. J Pediatr. 2018 May;196:168-174.e1. doi: 10.1016/j.jpeds.2018.01.028. Epub 2018 Mar 15. PMID 29551311
- [Derived] Sen S, Penfield-Cyr A, Hollis BW, Wagner CL. Maternal Obesity, 25-Hydroxy Vitamin D Concentration, and Bone Density in Breastfeeding Dyads. J Pediatr. 2017 Aug;187:147-152.e1. doi: 10.1016/j.jpeds.2017.04.024. Epub 2017 May 23. PMID 28549637
- [Derived] Hollis BW, Wagner CL, Howard CR, Ebeling M, Shary JR, Smith PG, Taylor SN, Morella K, Lawrence RA, Hulsey TC. Maternal Versus Infant Vitamin D Supplementation During Lactation: A Randomized Controlled Trial. Pediatrics. 2015 Oct;136(4):625-34. doi: 10.1542/peds.2015-1669. PMID 26416936

RESULTS

PARTICIPANT FLOW:
Groups:
- Control 400 IU Vitamin D3: 400 IU vitamin D3/day given to lactating women and 400 IU vitamin D3/day given as oral supplement to infant in dyad
  vitamin D3 (cholecalciferol): 400 IU vitamin D3/day given to lactating mother and 400 IU vitamin D3/day given to her infant
- 2400 IU Vitamin D3 (Cholecalciferol): 2400 IU vitamin D3 given to lactating mother: 400 IU vitamin D3 from a prenatal vitamin and 2000 IU vitamin D3 and 0 IU vitamin D3 (placebo) given to her breastfeeding infant
  Vitamin D3 (cholecalciferol): 2400 IU vitamin D3/day given to lactating women and 0 IU vitamin D3/day (placebo) given as oral supplement to her breastfeeding infant
- 6400 Vitamin D3 (Cholecalciferol): 6400 IU vitamin D3 given to lactating mother: 400 IU vitamin D3 from a prenatal vitamin and 6000 IU vitamin D3 and 0 IU vitamin D3 (placebo) given to her breastfeeding infant
  Vitamin D3 (cholecalciferol): 6400 IU vitamin D3/day given to lactating women and 0 IU vitamin D3/day (placebo) given as oral supplement to her breastfeeding infant
Period: Overall Study
Arm/Group | Control 400 IU Vitamin D3 | 2400 IU Vitamin D3 (Cholecalciferol) | 6400 Vitamin D3 (Cholecalciferol)
Started | 199 | 66 | 195
Completed | 122 | 44 | 128
Not Completed | 77 | 22 | 67

BASELINE CHARACTERISTICS:
Groups:
- 2400 Vitamin D3 (Cholecalciferol): 2400 IU vitamin D3 given to lactating mother: 400 IU vitamin D3 from a prenatal vitamin and 2000 IU vitamin D3 and 0 IU vitamin D3 (placebo) given to her breastfeeding infant
  Vitamin D3 (cholecalciferol): 2400 IU vitamin D3/day given to lactating women and 0 IU vitamin D3/day (placebo) given as oral supplement to her breastfeeding infant
- Total: Total of all reporting groups
Arm/Group | Control 400 IU Vitamin D3 | 2400 Vitamin D3 (Cholecalciferol) | 6400 Vitamin D3 (Cholecalciferol) | Total
Number analyzed (Participants) | 199 | 66 | 195 | 460
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 199 | 66 | 195 | 460
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.6 (6.2) | 29.4 (5.3) | 27.3 (5.9) | 27.7 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 66 | 195 | 460
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 199 | 66 | 195 | 460

OUTCOME MEASURES:

1. Primary Outcome: 25-Hydroxyvitamin D Levels for Postpartum Mother 7 Months After Delivery
Time Frame: to 7 months postpartum
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Control 400 IU Vitamin D3 | 2400 IU Vitamin D3 (Cholecalciferol) | 6400 Vitamin D3 (Cholecalciferol)
Number analyzed (Participants) | 122 | 44 | 128
ng/mL | 28.5 (11.5) | 38.0 (55.6) | 55.6 (23.4)

2. Secondary Outcome: Maternal Health Status - Vitamin D Deficiency
Description: Percentage of subjects with 25-hydroxyvitamin D [25(OH)D] concentration <20 ng/mL at Visit 7
Time Frame: to 7 months postpartum
Measure: Number; unit: percentage of participants
Arm/Group | Control 400 IU Vitamin D3 | 2400 IU Vitamin D3 (Cholecalciferol) | 6400 IU Vitamin D3 (Cholecalciferol)
Number analyzed (Participants) | 122 | 44 | 128
percentage of participants | 22.95 | 11.36 | 4.69

3. Secondary Outcome: Infant Health Status - Vitamin D Deficiency
Description: Percentage of infants with 25-hydroxyvitamin D [25(OH)D] concentration <20 ng/mL at Visit 7
Time Frame: to 7 months of age
Population: The number of infants analyzed in each group was fewer than the number of subjects analyzed for the maternal outcomes - though blood draws were attempted for all infants at Visit 7, we were unable to obtain blood from 14 infants in the 400 IU arm, 7 infants in the 2400 IU arm, and 14 infants in the 6400 IU arm.
Measure: Number; unit: percentage of infants
Arm/Group | Control 400 IU Vitamin D3 | 2400 IU Vitamin D3 (Cholecalciferol) | 6400 IU Vitamin D3 (Cholecalciferol)
Number analyzed (Participants) | 108 | 37 | 114
percentage of infants | 2.78 | 8.11 | 2.63

ADVERSE EVENTS:
Groups:
- 6400 IU Vitamin D3 (Cholecalciferol): 6400 IU vitamin D3 given to lactating mother: 400 IU vitamin D3 from a prenatal vitamin and 6000 IU vitamin D3 and 0 IU vitamin D3 (placebo) given to her breastfeeding infant
  Vitamin D3 (cholecalciferol): 6400 IU vitamin D3/day given to lactating women and 0 IU vitamin D3/day (placebo) given as oral supplement to her breastfeeding infant
Arm/Group | Control 400 IU Vitamin D3 | 2400 IU Vitamin D3 (Cholecalciferol) | 6400 IU Vitamin D3 (Cholecalciferol)
Serious Adverse Events (participants affected / at risk) | 2/199 | 0/66 | 1/195
Other Adverse Events (participants affected / at risk) | 11/199 | 6/66 | 8/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control 400 IU Vitamin D3 (N=199) | 2400 IU Vitamin D3 (Cholecalciferol) (N=66) | 6400 IU Vitamin D3 (Cholecalciferol) (N=195)
Sudden Unexpected Infant Death (General disorders) | 2 (2) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control 400 IU Vitamin D3 (N=199) | 2400 IU Vitamin D3 (Cholecalciferol) (N=66) | 6400 IU Vitamin D3 (Cholecalciferol) (N=195)
Postpartum complications within one year of delivery (General disorders) | 11 (11) | 6 (6) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No